CLINICAL TRIAL: NCT03582592
Title: Fluid Distribution Timetable on Adherence to Fluid Restriction of Patients With End-Stage Renal Disease Undergoing Hemodialysis: A Single-Blind, Randomized-Controlled Pilot Study
Brief Title: Fluid Distribution Timetable on Adherence to Fluid Restriction of Patients With End-Stage Renal Disease on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santo Tomas Hospital, Philippines (Other)
Responsible Party: Principal Investigator, Rame John L. Mina, Student Nurse, University of Santo Tomas Hospital, Philippines
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USTCON-2016-SR39
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: End-Stage Kidney Disease; Hemolysis; Nursing
Keywords: Fluid distribution timetable; Fluid restriction adherence; End-Stage Kidney Disease; Hemodialysis; Thirst; Interdialytic Weight Gain; Nursing
MeSH Terms: conditions — Kidney Failure, Chronic; Hemolysis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid Distribution Timetable (FDT) Group (Experimental): It is the fluid distribution timetable. It is a scheduled distribution of pre-determined amounts of fluid intake on a daily basis depicted via a 5x6 table. The timetable includes three major columns. The first column has six timepoints of a day with a four-hour interval. The second column, which was further divided into four sub-columns, reflects the percentage of fluid allotment for food, activities, medication, and thirst encounters. The percentage of fluid allocation was computed based on the patient's prescribed fluid restriction, usual time of food intakes in a day, usual level of activity, time of medication intake, and common time they encounter thirst in a day. Lastly, the third column indicates the converted percentages of fluid allotment in milliliters.
  Interventions: Behavioral: Fluid Distribution Timetable
- Comparison Group (No Intervention): It is the standard of care that served as the intervention. The control group received the standard care for patients on hemodialysis. The standard care involves a 10 -15-minute face-to-face health teaching of their treatment regimen including pharmacologic management, dialysis schedule, dietary and fluid restrictions or nutritional therapy, care for vascular access, and other necessary lifestyle modifications.

INTERVENTIONS:
Behavioral: Fluid Distribution Timetable — It is a scheduled distribution of pre-determined amounts of fluid intake on a daily basis depicted via a 5x6 table. The timetable includes three major columns. The first column has six timepoints of a day with a four-hour interval. The second column, which was further divided into four sub-columns, reflects the percentage of fluid allotment for food, activities, medication, and thirst encounters. The percentage of fluid allocation was computed based on the patient's prescribed fluid restriction, usual time of food intakes in a day, usual level of activity, time of medication intake, and common time they encounter thirst in a day. Lastly, the third column indicates the converted percentages of fluid allotment in milliliters.
  Arms: Fluid Distribution Timetable (FDT) Group

SUMMARY:
Fluid restriction is necessary among patients with chronic kidney disease. However, treatment adherence remains a challenge. Hence, this study determined the effects of a fluid distribution timetable on adherence to fluid restriction of patients with end-stage renal disease undergoing hemodialysis. This study used a single-blind, randomized-controlled pilot study design. Patients with end-stage renal disease were randomly-assigned using computer-generated sequences of randomly permuted blocks stratified according to sex to receive the fluid distribution timetable or standard care. Adherence to fluid restriction was measured using two indicators - thirst and interdialytic weight gain - and were compared using One-way RM-MANOVA and MANCOVA. Secondary outcomes included baseline patient demographic and clinical characteristics and were compared according to treatment allocation. Both groups were followed-up for four weeks, assessing outcome measures during the second hemodialysis session for each week.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD), defined as a condition in which the kidneys are damaged or cannot filter blood similar to a healthy kidney (Centers for Disease Control and Prevention, 2017), is a rising global dilemma. In fact, it has been a leading cause of morbidity and mortality worldwide, afflicting approximately 8% - 16% of the global population (Jha et al., 2013) and ranking eighth among the leading causes of death. It has also been acknowledged as a troublesome disorder causing a myriad of health-related problems (Lowney et al., 2015), financial burden (Bavanandan et al., 2016), and poor survival outcomes (Halle et al., 2016).

Hemodialysis, a form of renal replacement treatment, has been the mainstream management for patients with kidney diseases (Smeltzer et al., 2010) despite several health complications (Smeltzer et al., 2010; Lowney et al., 2015). However, dietary and fluid therapy are also necessary components of the management for patient with ESRD. A common concern among patients on hemodialysis is the non-adherence to fluid therapy. Although this management is simple, it remains a challenge to patients on hemodialysis because of several physiologic changes brought by ESRD. As a result, numerous problems such as fluid overload, electrolyte imbalances, and acid-base imbalances occur which are detrimental to the patient's overall health. Since patients on hemodialysis are the key players in promoting their health, it is, therefore, imperative to develop individualized and empowering strategies what will promote their adherence to fluid therapy. The proposed strategy in this study is the fluid distribution timetable, a simple and health promotive intervention involving scheduled distribution of pre-determined amounts of fluid intake on a daily basis. This intervention consider the various sources and usage of fluids per day and allocates fluid intake according to the patient's prescribed fluid restriction. Hence, this study determined the effects of a fluid distribution timetable on adherence to fluid restriction of patients with end-stage renal disease undergoing hemodialysis.

This study is a single-blind, single-center, randomized-controlled pilot study at the dialysis unit of a tertiary level government-owned institution in Quezon City, Philippines. Patients were randomly-allocated to receive fluid distribution timetable with standard care (intervention) or standard care alone (control). Random allocation of respondents was conducted using computer-generated sequences of randomly permuted blocks (sizes of three, four, and five) at our office. Randomization was carried out by an independent statistician and was stratified according to their sex. During the study period, treatment allocation was masked from site personnel and patients. Post-hoc power analysis for two group means, using GPower version 3.1, revealed that a sample size of 24 patients with a 1:1.20 group allocation ratio yields a power of 99% at a significance of 5% (two-sided) and detects an effect size of 0.80.

The control group received the standard care for patients on hemodialysis. The standard care involves a 10 -15-minute face-to-face health teaching of their treatment regimen including pharmacologic management, dialysis schedule, dietary and fluid restrictions or nutritional therapy, care for vascular access, and other necessary lifestyle modifications. The treatment group, on the other hand, received a combination of the standard care and the intervention, the fluid distribution timetable. It is a scheduled distribution of pre-determined amounts of fluid intake on a daily basis depicted via a 5x6 table. The timetable includes three major columns. The first column has six timepoints of a day with a four-hour interval. The second column, which was further divided into four sub-columns, reflects the percentage of fluid allotment for food, activities, medication, and thirst encounters. The percentage of fluid allocation was computed based on the patient's prescribed fluid restriction, usual time of food intakes in a day, usual level of activity, time of medication intake, and common time they encounter thirst in a day. Lastly, the third column indicates the converted percentages of fluid allotment in milliliters. In designing the intervention, we selected three behavior-specific cognitions from the Health Promotion Model by Nola J. Pender: perceived benefits, barriers, and self-efficacy. These cognitions are modifiable determinants of behavior that promote well-being. As such, the fluid distribution timetable enumerated the advantages of adherence and the disadvantages of non-adherence to fluid restriction.

Adherence to fluid restriction was measured using two indicators - thirst and interdialytic weight gain - and were compared using One-way RM-MANOVA and MANCOVA. Thirst was measured using a self-reported questionnaire the Dialysis Thirst Inventory, while interdialytic weight gain computed using a calibrated calculator by subtracting post-dialysis weight at the end of the previous hemodialysis session from the pre-dialysis weight during the current hemodialysis session. Secondary outcomes included baseline patient demographic and clinical characteristics and were compared according to treatment allocation. Both groups were followed-up for four weeks, assessing outcome measures during the second hemodialysis session for each week.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with end stage renal disease (ESRD);
* were oligoanuric (oliguria of <1mL/kg/hour or anuria over 6 hours);
* had been on hemodialysis for at least 6 months;
* were alert and oriented; and,
* were scheduled for hemodialysis twice a week

Exclusion Criteria:

* Patients who were pregnant;
* had a history of or has overt mental illness;
* were lethargic, disoriented, or debilitated during recruitment; and,
* had complicated medical conditions such as congestive heart failure and pulmonary congestion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived Thirst | 4 Weeks
  The Dialysis Thirst Inventory (DTI) measured perceived thirst among the participants. It is a 7-item questionnaire answered on 5-point Likert scale, with scores ranging from 7 to 35 and higher scores indicating higher thirst. No cut-off score is present for the questionnaire; however, higher scores are interpreted as higher perceived thirst.
Interdialytic Weight Gain | 4 Weeks
  It is the net increase in body weight from previous post-dialysis weight measured in kilograms

SECONDARY OUTCOMES:
Age | Week 1
  It refers to the age of the respondent in years at the time of participation in the study.
Sex | Week 1
  It refers to the biological gender assignment of the respondent at the time of participation in the study.
Educational Attainment | Week 1
  It refers to the highest educational attainment of the respondent and it is categorized into 5: no formal education, primary education, secondary education, college level, and post-graduate level.
Blood Pressure | 4 Weeks
  It refers to both the systolic and diastolic blood pressure, measured in mmHg, of the respondent.
Pulse Rate | 4 Weeks
  It refers to the number of heart beats per minute.
Respiratory Rate | 4 Weeks
  It refers to the number of respirations in minute of the respondent.
Edema Status | Week 1
  This refers to the edema status of the respondent at the time of participation in the study.
Ultrafiltration Goal | Week 1
  It refer to the ultrafiltration status of the respondent and it is categorized into to: met goal and unmet goal.

CONTACTS AND LOCATIONS:
Overall Officials: Rame John L Mina, BSN, RN, Principal Investigator — UST College of Nursing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mina RJL, Lerma MB, Litan PLB, Milano AAL, Mojica ADR, Malong-Consolacion CP, Lerma EB, Macindo JRB, Torres GCS. Fluid distribution timetable on adherence to fluid restriction of patients with end-stage renal disease undergoing haemodialysis: Single-blind, Randomized-Controlled Pilot Study. J Adv Nurs. 2019 Jun;75(6):1328-1337. doi: 10.1111/jan.13964. Epub 2019 Mar 18. PMID 30706521